CLINICAL TRIAL: NCT05257941
Title: Randomized Prospective Study Comparison of Erector Spinae Plane Block and Intrathecal Opioid for Postoperative Analgesia After Laparoscopic Colorectal Surgery in an Enhanced Recovery Setting
Brief Title: ESP Block VS Intrathecal Opioid After Laparoscopic Colorectal Surgery
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study specific patients are now scheduled at another hospital for this procedure
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Amy McCutchan, Assistant Professor of Clinical Anesthesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12514
Record Dates: First submitted 2022-01-25; First posted 2022-02-25 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IT Injection (Active Comparator): an intrathecal (IT) injection in the back in which a small dose duramorph and bupivacaine will be placed into the spinal fluid
  Interventions: Drug: IT Injection
- ESP Block (Active Comparator): an erector spinae plane (ESP) block in which bupivacaine and decadron are injected near the nerves under a muscle in the back.
  Interventions: Drug: ESP Block

INTERVENTIONS:
Drug: IT Injection — an intrathecal (IT) injection in the back in which a small dose duramorph and bupivacaine will be placed into the spinal fluid
  Arms: IT Injection
Drug: ESP Block — an erector spinae plane (ESP) block in which bupivacaine and decadron are injected near the nerves under a muscle in the back
  Arms: ESP Block

SUMMARY:
This study is being done to compare 2 types of pain control methods and determine which is more effective postoperatively for laparoscopic colorectal surgery. Group 1 will receive an intrathecal (IT) injection in the back in which a small dose duramorph and bupivacaine will be placed into the spinal fluid. Group 2 will receive an erector spinae plane (ESP) block in which bupivacaine and decadron are injected near the nerves under a muscle in the back.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective laparoscopic colorectal procedure at Indiana University Hospital or Methodist Hospital
* ASA Class 1, 2, 3 (American Society of Anesthesiologists physical status classification system)
* Age 18 to 80 years (male or female)
* BMI < 40kg/m2
* Desires regional anesthesia for postoperative pain control

Exclusion Criteria:

* Any contraindication for neuraxial analgesia or ESP block procedure

  * Contraindications for neuraxial analgesia include: Elevated intracranial pressure (except in cases of pseudo-tumor cerebri), infection at the site of injection, lack of consent from the patient, patient refusal, true allergy to any drug used in the spine, and uncorrected hypovolemia.
  * Contraindications for ESP block procedure include: Infection at the site of injection, patient refusal, true allergy to any of the drugs used in the block, and lack of patient consent.
* Any patient undergoing a laparoscopic abdominoperineal resection.
* Any physical, mental or medical conditions which, in the opinion of the investigators, may confound quantifying postoperative pain resulting from surgery.
* Known true allergy to the study medications (morphine, bupivacaine, decadron, Tylenol, Celebrex)
* Takes over 30 mg of oral morphine equivalents daily
* Any history of substance abuse in the past 6 months
* End stage liver disease, end stage renal disease
* Body weight of < 50 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
cumulated oral morphine equivalent (OME) | 24 hours after surgery
  morphine consumption

SECONDARY OUTCOMES:
opioid consumption | 1 hour after surgery
  opioid consumption in OME
opioid consumption | 12 hours after surgery
  opioid consumption in OME
opioid consumption | 24 hours after surgery
  opioid consumption in OME
opioid consumption | 48 hours after surgery
  opioid consumption in OME
opioid consumption | 72 hours after surgery
  opioid consumption in OME
Visual Analog Scale pain scores | 1 hour after surgery
  pain scores using the Visual Analog Scale (0-10 with 0 being no pain and 10 being the worst pain)
Visual Analog Scale pain scores | 12 hours after surgery
  pain scores using the Visual Analog Scale (0-10 with 0 being no pain and 10 being the worst pain)
Visual Analog Scale pain scores | 24 hours after surgery
  pain scores using the Visual Analog Scale (0-10 with 0 being no pain and 10 being the worst pain)
Visual Analog Scale pain scores | 48 hours after surgery
  pain scores using the Visual Analog Scale (0-10 with 0 being no pain and 10 being the worst pain)
Visual Analog Scale pain scores | 72 hours after surgery
  pain scores using the Visual Analog Scale (0-10 with 0 being no pain and 10 being the worst pain)
opioid side effects | duration of hospital stay up to 72 hours
  incidence of opioid side effects (nausea, pruritus, urinary retention, respiratory depression, ileus)
first ambulation | duration of hospital stay up to 72 hours
  time to patient first ambulation
first flatus | duration of hospital stay up to 72 hours
  time to first flatus
oral liquid | duration of hospital stay up to 72 hours
  time to first oral liquid intake
oral food | duration of hospital stay up to 72 hours
  time to first oral food intake
hospital stay | duration of hospital stay up to 7 days
  amount of time each subject spends in the hospital before discharge
patient's satisfaction scores | 24 hours after surgery
  assess patient's satisfaction with care (1-10 with 1 being the least satisfied and 10 being the most satisfied)
patient's satisfaction scores | 48 hours after surgery
  assess patient's satisfaction with care (1-10 with 1 being the least satisfied and 10 being the most satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Amy McCutchan, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- IU Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kehlet H, Wilmore DW. Evidence-based surgical care and the evolution of fast-track surgery. Ann Surg. 2008 Aug;248(2):189-98. doi: 10.1097/SLA.0b013e31817f2c1a. PMID 18650627
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Miller TE, Thacker JK, White WD, Mantyh C, Migaly J, Jin J, Roche AM, Eisenstein EL, Edwards R, Anstrom KJ, Moon RE, Gan TJ; Enhanced Recovery Study Group. Reduced length of hospital stay in colorectal surgery after implementation of an enhanced recovery protocol. Anesth Analg. 2014 May;118(5):1052-61. doi: 10.1213/ANE.0000000000000206. PMID 24781574
- [Background] Wind J, Polle SW, Fung Kon Jin PH, Dejong CH, von Meyenfeldt MF, Ubbink DT, Gouma DJ, Bemelman WA; Laparoscopy and/or Fast Track Multimodal Management Versus Standard Care (LAFA) Study Group; Enhanced Recovery after Surgery (ERAS) Group. Systematic review of enhanced recovery programmes in colonic surgery. Br J Surg. 2006 Jul;93(7):800-9. doi: 10.1002/bjs.5384. PMID 16775831
- [Background] Lassen K, Soop M, Nygren J, Cox PB, Hendry PO, Spies C, von Meyenfeldt MF, Fearon KC, Revhaug A, Norderval S, Ljungqvist O, Lobo DN, Dejong CH; Enhanced Recovery After Surgery (ERAS) Group. Consensus review of optimal perioperative care in colorectal surgery: Enhanced Recovery After Surgery (ERAS) Group recommendations. Arch Surg. 2009 Oct;144(10):961-9. doi: 10.1001/archsurg.2009.170. PMID 19841366
- [Background] Khoo CK, Vickery CJ, Forsyth N, Vinall NS, Eyre-Brook IA. A prospective randomized controlled trial of multimodal perioperative management protocol in patients undergoing elective colorectal resection for cancer. Ann Surg. 2007 Jun;245(6):867-72. doi: 10.1097/01.sla.0000259219.08209.36. PMID 17522511
- [Background] McEvoy MD, Scott MJ, Gordon DB, Grant SA, Thacker JKM, Wu CL, Gan TJ, Mythen MG, Shaw AD, Miller TE; Perioperative Quality Initiative (POQI) I Workgroup. American Society for Enhanced Recovery (ASER) and Perioperative Quality Initiative (POQI) joint consensus statement on optimal analgesia within an enhanced recovery pathway for colorectal surgery: part 1-from the preoperative period to PACU. Perioper Med (Lond). 2017 Apr 13;6:8. doi: 10.1186/s13741-017-0064-5. eCollection 2017. PMID 28413629
- [Background] Marret E, Remy C, Bonnet F; Postoperative Pain Forum Group. Meta-analysis of epidural analgesia versus parenteral opioid analgesia after colorectal surgery. Br J Surg. 2007 Jun;94(6):665-73. doi: 10.1002/bjs.5825. PMID 17514701
- [Background] Borzellino G, Francis NK, Chapuis O, Krastinova E, Dyevre V, Genna M. Role of Epidural Analgesia within an ERAS Program after Laparoscopic Colorectal Surgery: A Review and Meta-Analysis of Randomised Controlled Studies. Surg Res Pract. 2016;2016:7543684. doi: 10.1155/2016/7543684. Epub 2016 Aug 24. PMID 27642630
- [Background] Liu H, Hu X, Duan X, Wu J. Thoracic epidural analgesia (TEA) vs. patient controlled analgesia (PCA) in laparoscopic colectomy: a meta-analysis. Hepatogastroenterology. 2014 Jul-Aug;61(133):1213-9. PMID 25436285
- [Background] Merchea A, Lovely JK, Jacob AK, Colibaseanu DT, Kelley SR, Mathis KL, Spears GM, Huebner M, Larson DW. Efficacy and Outcomes of Intrathecal Analgesia as Part of an Enhanced Recovery Pathway in Colon and Rectal Surgical Patients. Surg Res Pract. 2018 Mar 1;2018:8174579. doi: 10.1155/2018/8174579. eCollection 2018. PMID 29687077
- [Background] Koning MV, Klimek M, Rijs K, Stolker RJ, Heesen MA. Intrathecal hydrophilic opioids for abdominal surgery: a meta-analysis, meta-regression, and trial sequential analysis. Br J Anaesth. 2020 Sep;125(3):358-372. doi: 10.1016/j.bja.2020.05.061. Epub 2020 Jul 11. PMID 32660719
- [Background] Day AR, Smith RV, Scott MJ, Fawcett WJ, Rockall TA. Randomized clinical trial investigating the stress response from two different methods of analgesia after laparoscopic colorectal surgery. Br J Surg. 2015 Nov;102(12):1473-9. doi: 10.1002/bjs.9936. Epub 2015 Sep 23. PMID 26395762
- [Background] Levy BF, Scott MJ, Fawcett W, Fry C, Rockall TA. Randomized clinical trial of epidural, spinal or patient-controlled analgesia for patients undergoing laparoscopic colorectal surgery. Br J Surg. 2011 Aug;98(8):1068-78. doi: 10.1002/bjs.7545. Epub 2011 May 17. PMID 21590762
- [Background] Pedrazzani C, Menestrina N, Moro M, Brazzo G, Mantovani G, Polati E, Guglielmi A. Local wound infiltration plus transversus abdominis plane (TAP) block versus local wound infiltration in laparoscopic colorectal surgery and ERAS program. Surg Endosc. 2016 Nov;30(11):5117-5125. doi: 10.1007/s00464-016-4862-5. Epub 2016 Mar 22. PMID 27005290
- [Background] Liu X, Song T, Chen X, Zhang J, Shan C, Chang L, Xu H. Quadratus lumborum block versus transversus abdominis plane block for postoperative analgesia in patients undergoing abdominal surgeries: a systematic review and meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 Mar 2;20(1):53. doi: 10.1186/s12871-020-00967-2. PMID 32122319
- [Background] Dam M, Hansen C, Poulsen TD, Azawi NH, Laier GH, Wolmarans M, Chan V, Bendtsen TF, Borglum J. Transmuscular quadratus lumborum block reduces opioid consumption and prolongs time to first opioid demand after laparoscopic nephrectomy. Reg Anesth Pain Med. 2021 Jan;46(1):18-24. doi: 10.1136/rapm-2020-101745. Epub 2020 Oct 26. PMID 33106280
- [Background] Huang J, Liu JC. Ultrasound-guided erector spinae plane block for postoperative analgesia: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 Apr 14;20(1):83. doi: 10.1186/s12871-020-00999-8. PMID 32290814
- [Background] Kendall MC, Alves L, Traill LL, De Oliveira GS. The effect of ultrasound-guided erector spinae plane block on postsurgical pain: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 May 1;20(1):99. doi: 10.1186/s12871-020-01016-8. PMID 32357842
- [Background] Kwon HM, Kim DH, Jeong SM, Choi KT, Park S, Kwon HJ, Lee JH. Does Erector Spinae Plane Block Have a Visceral Analgesic Effect?: A Randomized Controlled Trial. Sci Rep. 2020 May 21;10(1):8389. doi: 10.1038/s41598-020-65172-0. PMID 32439926
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] López MB, Cadórniga ÁG, González JML, Suárez ED, Carballo CL, Sobrino FP. Erector spinae block. A narrative review. Cent Eur J Clin Res. 2018;1(1):28-39
- [Background] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] Tulgar S, Ahiskalioglu A, De Cassai A, Gurkan Y. Efficacy of bilateral erector spinae plane block in the management of pain: current insights. J Pain Res. 2019 Aug 27;12:2597-2613. doi: 10.2147/JPR.S182128. eCollection 2019. PMID 31695476
- [Background] Hamed MA, Goda AS, Basiony MM, Fargaly OS, Abdelhady MA. Erector spinae plane block for postoperative analgesia in patients undergoing total abdominal hysterectomy: a randomized controlled study original study. J Pain Res. 2019 Apr 30;12:1393-1398. doi: 10.2147/JPR.S196501. eCollection 2019. PMID 31118757
- [Background] Rashid A, Gorissen KJ, Ris F, Gosselink MP, Shorthouse JR, Smith AD, Pandit JJ, Lindsey I, Crabtree NA. No benefit of ultrasound-guided transversus abdominis plane blocks over wound infiltration with local anaesthetic in elective laparoscopic colonic surgery: results of a double-blind randomized controlled trial. Colorectal Dis. 2017 Jul;19(7):681-689. doi: 10.1111/codi.13578. PMID 27943522
- [Background] Oh TK, Yim J, Kim J, Eom W, Lee SA, Park SC, Oh JH, Park JW, Park B, Kim DH. Effects of preoperative ultrasound-guided transversus abdominis plane block on pain after laparoscopic surgery for colorectal cancer: a double-blind randomized controlled trial. Surg Endosc. 2017 Jan;31(1):127-134. doi: 10.1007/s00464-016-4941-7. Epub 2016 Apr 29. PMID 27129571
- [Background] Dewinter G, Coppens S, Van de Velde M, D'Hoore A, Wolthuis A, Cuypers E, Rex S. Quadratus Lumborum Block Versus Perioperative Intravenous Lidocaine for Postoperative Pain Control in Patients Undergoing Laparoscopic Colorectal Surgery: A Prospective, Randomized, Double-blind Controlled Clinical Trial. Ann Surg. 2018 Nov;268(5):769-775. doi: 10.1097/SLA.0000000000002888. PMID 30004914
- [Background] Boulianne M, Paquet P, Veilleux R, Drolet S, Meunier A, Frigault J, Simonyan D, Turgeon AF. Effects of quadratus lumborum block regional anesthesia on postoperative pain after colorectal resection: a randomized controlled trial. Surg Endosc. 2020 Sep;34(9):4157-4165. doi: 10.1007/s00464-019-07184-0. Epub 2019 Oct 22. PMID 31641913
- [Background] Koo CH, Hwang JY, Shin HJ, Ryu JH. The Effects of Erector Spinae Plane Block in Terms of Postoperative Analgesia in Patients Undergoing Laparoscopic Cholecystectomy: A Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2020 Sep 10;9(9):2928. doi: 10.3390/jcm9092928. PMID 32927867
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392
- [Background] Aksu C, Kuş A, Yörükoğlu HU, Tor Kılıç C, Gürkan Y. The effect of erector spinae plane block on postoperative pain following laparoscopic cholecystectomy: a randomized controlled study. JARSS 2019;27(1):9-14
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Schwartzmann A, Peng P, Maciel MA, Alcarraz P, Gonzalez X, Forero M. A magnetic resonance imaging study of local anesthetic spread in patients receiving an erector spinae plane block. Can J Anaesth. 2020 Aug;67(8):942-948. doi: 10.1007/s12630-020-01613-8. Epub 2020 Mar 9. PMID 32152885
- [Background] Vidal E, Gimenez H, Forero M, Fajardo M. Erector spinae plane block: A cadaver study to determine its mechanism of action. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Nov;65(9):514-519. doi: 10.1016/j.redar.2018.07.004. Epub 2018 Aug 27. English, Spanish. PMID 30166123
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Kamel AAF, Amin OAI, Ibrahem MAM. Bilateral Ultrasound-Guided Erector Spinae Plane Block Versus Transversus Abdominis Plane Block on Postoperative Analgesia after Total Abdominal Hysterectomy. Pain Physician. 2020 Jul;23(4):375-382. PMID 32709172
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT05257941/Prot_SAP_000.pdf